CLINICAL TRIAL: NCT03061981
Title: A Phase I, First In Human, Double Blind, Placebo Controlled, Single Ascending Dose Study To Evaluate The Safety, Tolerability, Pharmacokinetics, Pharmacodynamics And Interaction Effect With Metformin Following A Single Oral Dose Of DA-1241 In Healthy Male Subjects
Brief Title: A Study To Evaluate The Safety,Tolerability, PK and PD Of DA-1241 In Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1241_DM_Ia
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; DA-1241

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DA-1241:8 subjects in each cohort(Cohort 1-6) (Active Comparator): Subjects will participate in 1 of 6 cohorts consisting of 10 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 8:2 (DA-1241 to matching placebo).
  Interventions: Drug: DA-1241
- Placebo: 2 subjects in each cohort(Cohort 1-6) (Placebo Comparator): Subjects will participate in 1 of 6 cohorts consisting of 10 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 8:2 (DA-1241 to matching placebo).
  Interventions: Drug: Placebo
- DA-1241 in IE Cohort: 8 subjects in choosen cohort (Other): One of the cohorts will be selected,based on a review of the data from cohort 1-6, to assess the IE of metformin on the PK of DA-1241.
  Interventions: Drug: Metformin; Drug: DA-1241
- Placebo in IE Cohort: 2 subjects in choosen cohort (Other): One of the cohorts will be selected,based on a review of the data from cohort 1-6, to assess the IE of metformin on the PK of DA-1241.
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: Placebo — After pre-dose assessments on Day 1, subjects will receive a single oral dose of IMP after an overnight fast in each Treatment Period.
  Arms: Placebo in IE Cohort: 2 subjects in choosen cohort; Placebo: 2 subjects in each cohort(Cohort 1-6)
Drug: Metformin — Subjects in the IE cohort will receive 500 mg metformin (IR formulation) at 12 hours on Day 1 and a single oral dose of the IMP with 500 mg metformin (IR formulation) after an overnight fast on Day 1, in Treatment Period 2.
  Arms: DA-1241 in IE Cohort: 8 subjects in choosen cohort; Placebo in IE Cohort: 2 subjects in choosen cohort
Drug: DA-1241 — After pre-dose assessments on Day 1, subjects will receive a single oral dose of IMP after an overnight fast in each Treatment Period .
  Arms: DA-1241 in IE Cohort: 8 subjects in choosen cohort; DA-1241:8 subjects in each cohort(Cohort 1-6)

SUMMARY:
This is a randomized, double blind, placebo controlled, single ascending dose study to assess the safety, tolerability, PK, PD and IE with metformin following a single oral dose of DA-1241 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent before any of the screening procedures are performed.
2. Male subjects aged between 18 and 55 years (both inclusive) at screening.
3. Body mass index (BMI) of 18.5 to 32.0 kg/m2 (both inclusive) at screening.
4. Medical history, vital signs, physical examination, standard 12-lead ECGs and laboratory investigations (clinical chemistry, hematology and urinalysis) must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the PI considers the deviation to be irrelevant for the purpose of the study. These assessments may be repeated once at the discretion of the PI.
5. Subjects with partners of childbearing potential must be willing to use medically acceptable double barrier forms of contraception from IMP administration until at least 3 months after the last day of IMP administration. Subjects must not donate sperm for the duration of the study and for at least 3 months after the last day of IMP administration.
6. Is a non-smoker or non-tobacco/nicotine user confirmed with urine cotinine test at screening and on admission to the EPCU. Nicotine products include, but are not limited to, tobacco cigarettes, electronic cigarettes, snuff, cigars, and pipes, including hookah or water pipes. The use of nicotine patches or gum (e.g., products used as part of a smoking cessation program) is not allowed.

Exclusion Criteria:

1. Has a known hypersensitivity to any component of the formulation of DA- 1241 or any of the excipients or to medicinal products with similar chemical structures.
2. Has a history or presence of any clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal or endocrine disease or other abnormality that may impact the ability of the subject to participate or potentially confound the study results.
3. Has a glycated hemoglobin A1C (HgbA1C) of ≥ 6.5% consistent with possible diabetes at screening.
4. Any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
5. Any concurrent disease or condition that, in the opinion of the PI, would make the subject unsuitable for participation in the clinical study.
6. Subject has a history of drinking > 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the EPCU.
7. Have positive test results for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibodies (anti HCV) or human immunodeficiency virus 1 and/or -2 antibodies (anti HIV-1 and/or -2) at screening.
8. History of drug abuse or has a positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, etc.) at screening or on Day 1.
9. Has donated or lost 450 mL or more of his blood volume (including plasmaphoresis), or had a transfusion of any blood product within 3 months before screening.
10. Taking any medication including prescription, herbal remedies, vitamin supplements, dietary supplements or other over-the-counter (OTC) products within 14 days or 5 half-lives of the product (whichever period is longer) before admission to the EPCU.
11. Has an abnormal (clinically significant) ECG at screening or on Day 1. Entry of any subject with an abnormal (but not clinically significant) ECG must be approved and documented by signature, by the PI or medically qualified Sub-investigator.
12. Has a supine blood pressure (BP) outside the ranges of 90 to 140 mmHg, inclusive, for systolic BP and 50 to 90 mmHg, inclusive, for diastolic BP, or has a resting heart rate outside the range of 45 to 100 beats per minute (bpm). If any of the values are out of range, the assessment may be repeated once for eligibility determination, at screening and admission on Day 1.
13. Has a corrected QT interval using Fridericia's corrected formula (QTcF) interval greater than 450 msec or PR interval outside the range of 120 to 220 msec. If any values are out of range, the ECG may be repeated once for eligibility determination, at screening and admission on Day 1.
14. Has an abnormal laboratory value that suggests a clinically significant underlying disease or has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values greater than 1.5 times the upper limit of normal (ULN). Laboratory assessments may be repeated once to confirm eligibility at screening and on Day 1.
15. Participation in another study with an experimental drug within 30 days or 5 half-lives, whichever is longer, of this study's screening visit. Participation is defined as the date of last dose received in the previous study.
16. Unwilling to abstain from vigorous exercise within 48 hours before Day 1.
17. Intake of any food or drinks containing grapefruit, Chinese grapefruit (pomelo), star fruit, pomegranate or Seville orange (including marmalade) within 48 hours before admission to the EPCU.
18. Have used alcohol within 72 hours prior to screening or within 72 hours prior to admission to the EPCU.
19. Is unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.
20. Is a study-site employee or an immediate family member or dependent (e.g., spouse, parent, child or sibling) of a study-site employee who is involved in the conduct of this study.
21. Has difficulty swallowing 2 tablets at the same time.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
[Safety and Tolerability] 12-lead ECGs, Vital signs. Physical examinations, Clinical laboratory testing and Adverse event assessments | Through study completion, an average of 40 days for each treatment period

SECONDARY OUTCOMES:
Maximum concentration of DA-1241 (Cmax) | Through the treatment period; 72 hours
Time of maximum plasma DA-1241 concentration (Tmax) | Through the treatment period; 72 hours
Area under the concentration-time curve (AUC) | Through the treatment period; 72 hours
Apparent terminal elimination half-life (t½) | Through the treatment period; 72 hours
Apparent total systemic clearance after oral administration (CL/F) | Through the treatment period; 72 hours
Apparent volume of distribution (Vz/F) | Through the treatment period; 72 hours
Amount of DA-1241 excreted unchanged in the urine in each collection interval(Ae) | Through the treatment period; 72 hours
Cumulative amount of DA-1241 excreted unchanged in the urine (Cum Ae) | Through the treatment period; 72 hours
Percentage fraction of DA-1241 excreted unchanged in the urine in each collection interval(Fe) | Through the treatment period; 72 hours
Cumulative percentage fraction of DA-1241 excreted unchanged in the urine (Cum Fe) | Through the treatment period; 72 hours
Renal clearance (CLR) | Through the treatment period; 72 hours

OTHER OUTCOMES:
Key metabolites of DA-1241 in Cohort 6 | Through the treatment period; 264 hours
  Blood samples and urine samples taken for PK (or PD) analysis will be used. Metabolites to be measured are not determined yet.

CONTACTS AND LOCATIONS:
Locations (1):
- Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No